CLINICAL TRIAL: NCT06544681
Title: Evaluation and Treatment Strategy Development of Coronary Heart Disease Guided by Optical Coherence Tomography Based on Multimodal Deep Learning
Brief Title: Evaluation and Treatment Strategy Development of Coronary Heart Disease Guided by OCT Based on Multimodal Deep Learning
Status: Not yet recruiting | Type: Observational
Sponsor: Xiang Ma (Other)
Collaborators: Shihezi University (Other)
Responsible Party: Sponsor-Investigator, Xiang Ma, professor, First Affiliated Hospital of Xinjiang Medical University
Organization: First Affiliated Hospital of Xinjiang Medical University (Other)
Other Study IDs: 2022B03022-3
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Coronary Disease; Coronary Artery Disease
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Coronary Stent Malapposition: Measurement results of deep learning-based OCT system: Coronary Stent Malapposition
  Interventions: Procedure: Coronary stenting with planned drug eluting stent (DES).
- Coronary Stent Well Apposed: Measurement results of a deep learning-based OCT system: Coronary Stent Well Apposed
  Interventions: Procedure: Coronary stenting with planned drug eluting stent (DES).

INTERVENTIONS:
Procedure: Coronary stenting with planned drug eluting stent (DES). — Stenting will be performed with OCT guidance according to the algorithm described in the protocol. A deep learning-based OCT system was used to measure the adherence of coronary stents.

SUMMARY:
This is a retrospective, multicenter, observational study aimed at assessing stent apposition for coronary stent implantation by an optical coherence tomography system constructed by deep learning algorithms and evaluating the prognosis of patients after stent implantation in conjunction with multimodal diagnostic and therapeutic information.

DETAILED DESCRIPTION:
In this study, we planned to retrospectively collect 2,000 subjects who underwent optical coherence tomography-guided percutaneous coronary stent implantation with an optical coherence tomography system constructed by a deep learning algorithm from 3 centers to assess stent apposition for coronary stent implantation, and to classify subjects into a group with poor stent apposition (axial distance >400 μm or length >1 mm) and a group with good stent apposition. All subjects were followed up within 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old;
* Angiography was performed, and OCT imaging of criminal blood vessels was performed before intervention;
* Type of coronary heart disease: Unstable angina pectoris (UA), ST elevation myocardial infarction (STEMI) And non-ST elevation myocardial infarction (NSTEMI);

Exclusion Criteria:

* Lack of medical records;
* Failure to complete follow-up;
* Previous coronary artery bypass grafting;
* Severe liver or kidney insufficiency;
* Infectious diseases, malignancies and bleeding diseases;
* OCT image quality was caused by large thrombus volume or residual blood in lumen and percutaneous coronary angiography Poor and further excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective data were collected from the First Affiliated Hospital of Xinjiang Medical University and Jining, Shandong Province from 2015 to 2022 Coronary artery disease patients undergoing coronary angiography and OCT examination in the First People's Hospital of China and Xigu District People's Hospital of Gansu Province.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | Post-procedure within 1 year
  Patients were followed up within 1 year after OCT and PCI. The follow-up included major adverse cardiac events: All causes were death, recurrent myocardial infarction, target vessel reconstruction, and stent thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Pengfei Liu, M.D, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Xinliang Peng, M.D, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Abudusalamu Tuerdimaimaiti, M.D, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University